CLINICAL TRIAL: NCT06116591
Title: A Phase 2, Randomized, Open-Label Trial to Describe the Safety and Immunogenicity of a Monovalent Pneumococcal Conjugate Candidate Administered As a 2-Dose Series in Healthy Toddlers 11 Through 15 Months of Age Who Previously Received the PCV10 Primary Series
Brief Title: A Phase 2 Study to Learn About a Monovalent Pneumococcal Conjugate Candidate in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C4801002; 2023-505154-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPnC candidate (Experimental): Participants will receive the mPnC candidate at Visit 1 and Visit 3 (approximately 8 weeks apart). PCV10 will also be given at Visit 1.
  Interventions: Biological: mPnC candidate
- mPnC control (Active Comparator): Participants will receive the mPnC control at Visit 1 and Visit 3 (approximately 8 weeks apart). PCV10 will also be given at Visit 1.
  Interventions: Biological: mPnC control

INTERVENTIONS:
Biological: mPnC candidate — monovalent pneumococcal conjugate candidate
  Arms: mPnC candidate
Biological: mPnC control — monovalent pneumococcal conjugate control
  Arms: mPnC control

SUMMARY:
The purpose of the study is to learn about the effects of a monovalent (single component) pneumococcal conjugate candidate (mPnC candidate) when given to toddlers between 11 and 15 months of age.

All participants in this study will receive 2 doses of either mPnC candidate or mPnC control at the clinic approximately 8 weeks apart. All participants will also receive their third (toddler) dose of PCV10 at Visit 1.

ELIGIBILITY:
Key Inclusion Criteria:

* Toddlers ≥11 to ≤15 months of age at the time of consent.
* Have received exactly 2 infant doses of PCV10 according to a local immunization schedule.
* Healthy toddlers determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Key Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of study intervention, 13vPnC, 20vPnC, or any diphtheria toxoid-containing vaccine.
* significant neurological disorder or history of seizure (excluding febrile seizure) or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders.
* Major known congenital malformation or serious chronic disorder.
* History of microbiologically proven invasive disease caused by S pneumoniae.
* Previous vaccination with any licensed pneumococcal vaccine (other than the PCV10 primary infant series) or investigational pneumococcal vaccine, or planned receipt of nonstudy pneumococcal vaccine during study participation.

Ages: 11 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Finland (9):
  - FVR, Kokkolan rokotetutkimusklinikka, Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka, Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka, Tampere, Pirkanmaa
  - FVR, Seinäjoen rokotetutkimusklinikka, Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka, Turku, Southwest Finland
  - FVR, Espoon rokotetutkimusklinikka, Espoo, Uusimaa
  - FVR, Etelä-Helsingin rokotetutkimusklinikka, Helsinki, Uusimaa
  - MeVac - Meilahti Vaccine Research Center, Helsinki, Uusimaa
  - FVR, Järvenpään rokotetutkimusklinikka, Jarvenpaa, Uusimaa
- Poland (2):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - NZOZ Praktyka Lekarza Rodzinnego "ESKULAP", Lublin, Lublin Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4801002

RESULTS

PARTICIPANT FLOW:
Groups:
- mPnC Candidate: Participants who had previously received 2 doses of 10-valent pneumococcal conjugate vaccine (PCV10) primary series as part of their infant routine vaccines were administered 0.5 milliliter (mL) dose of monovalent pneumococcal conjugate (mPnC) candidate intramuscularly at Visit 1 of the study (Day 1 of study; Dose 1) and Visit 3 of the study (56 to 70 days after Visit 1; Dose 2). Participants also received their third (toddler) dose of PCV10 at Visit 1 per childhood vaccine standard of care.
- mPnC Control: Participants who had previously received 2 doses of PCV10 primary series as part of their infant routine vaccines were administered 0.5 mL dose of mPnC control intramuscularly at Visit 1 of the study (Day 1 of study; Dose 1) and Visit 3 of the study (56 to 70 days after Visit 1; Dose 2). Participants also received their third (toddler) dose of PCV10 at Visit 1 per childhood vaccine standard of care.
Period: Overall Study
Arm/Group | mPnC Candidate | mPnC Control
Started | 52 | 53
Dose 1 at Study Visit 1 | 52 | 53
Dose 2 at Study Visit 3 | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 2
Not completed — No longer met eligibility criteria | 0 | 1
Not completed — Other: Change in life situation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- mPnC Candidate: Participants who had previously received 2 doses of PCV10 primary series as part of their infant routine vaccines were administered 0.5 mL dose of mPnC candidate intramuscularly at Visit 1 of the study (Day 1 of study; Dose 1) and Visit 3 of the study (56 to 70 days after Visit 1; Dose 2). Participants also received their third (toddler) dose of PCV10 at Visit 1 per childhood vaccine standard of care.
- Total: Total of all reporting groups
Arm/Group | mPnC Candidate | mPnC Control | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: Months] | 11.4 (0.56) | 11.3 (0.54) | 11.3 (0.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 25 | 28 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 52 | 51 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1
Description: Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild: > 0 to 2.0 centimeter (cm), moderate: >2.0 to 7.0 cm, severe: >7.0 cm and Grade 4: necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild: hurt if gently touched, moderate: hurt if gently touched, with crying, severe: caused limitation of limb movement and Grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain at injection site. Grade 4 assessments were made by the investigator. Any local reaction: any mild, moderate, severe, or Grade 4 redness, swelling, or pain at the injection site.
Time Frame: Day 1 through Day 7, where Day 1 is the day of Dose 1 administration (Visit 1 of study)
Population: Safety analysis set included all participants who received at least 1 dose of the study intervention. Here, ''Overall Number of Participants Analyzed'' signifies participants who received Dose 1 and who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 53
Percentage of participants
  Redness: Any | 17.3 [8.2 to 30.3] | 15.1 [6.7 to 27.6]
  Redness: Mild | 17.3 [8.2 to 30.3] | 9.4 [3.1 to 20.7]
  Redness: Moderate | 0 [0.0 to 6.8] | 5.7 [1.2 to 15.7]
  Redness: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Redness: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Swelling: Any | 15.4 [6.9 to 28.1] | 7.5 [2.1 to 18.2]
  Swelling: Mild | 11.5 [4.4 to 23.4] | 5.7 [1.2 to 15.7]
  Swelling: Moderate | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.1]
  Swelling: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Swelling: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Pain at the injection site: Any | 28.8 [17.1 to 43.1] | 30.2 [18.3 to 44.3]
  Pain at the injection site: Mild | 21.2 [11.1 to 34.7] | 17.0 [8.1 to 29.8]
  Pain at the injection site: Moderate | 5.8 [1.2 to 15.9] | 13.2 [5.5 to 25.3]
  Pain at the injection site: Severe | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.7]
  Pain at the injection site: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild: > 0 to 2.0 cm, moderate: >2.0 to 7.0 cm, severe: >7.0 cm and Grade 4: necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild: hurt if gently touched, moderate: hurt if gently touched, with crying, severe: caused limitation of limb movement and Grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain at injection site. Grade 4 assessments were made by the investigator. Any local reaction: any mild, moderate, severe, or Grade 4 redness, swelling, or pain at the injection site.
Time Frame: Day 1 through Day 7, where Day 1 is the day of Dose 2 administration (Visit 3 of study)
Population: Safety analysis set included all participants who received at least 1 dose of the study intervention. Here, ''Overall Number of Participants Analyzed'' signifies participants who received Dose 2 and who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 51
Percentage of participants
  Redness: Any | 13.5 [5.6 to 25.8] | 17.6 [8.4 to 30.9]
  Redness: Mild | 9.6 [3.2 to 21.0] | 15.7 [7.0 to 28.6]
  Redness: Moderate | 3.8 [0.5 to 13.2] | 2.0 [0.0 to 10.4]
  Redness: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Redness: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Swelling: Any | 0 [0.0 to 6.8] | 7.8 [2.2 to 18.9]
  Swelling: Mild | 0 [0.0 to 6.8] | 7.8 [2.2 to 18.9]
  Swelling: Moderate | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Swelling: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Swelling: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Pain at the injection site: Any | 15.4 [6.9 to 28.1] | 17.6 [8.4 to 30.9]
  Pain at the injection site: Mild | 11.5 [4.4 to 23.4] | 11.8 [4.4 to 23.9]
  Pain at the injection site: Moderate | 3.8 [0.5 to 13.2] | 5.9 [1.2 to 16.2]
  Pain at the injection site: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Pain at the injection site: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]

3. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Fever (oral temperature >= 38 degree Celsius [degC]) was categorized as >=38.0-38.4 degC, >38.4-38.9 degC, >38.9-40.0 degC and >40.0 degC. Decreased appetite was graded as mild: decreased interest in eating, moderate: decreased oral intake, severe: refusal to feed. Drowsiness was graded as mild: increased/prolonged sleeping bouts, moderate: slightly subdued, interfered daily activity, severe: disabled, not interested in daily activity. Irritability was graded as mild: easily consolable, moderate: required increased attention, severe: inconsolable, crying couldn't be comforted. Grade 4 decreased appetite, drowsiness and irritability events led to emergency room visit or hospitalization and were classified by investigator/medically qualified person. Any systemic event: any fever, decreased appetite, drowsiness, irritability.
Time Frame: Day 1 through Day 7, where Day 1 is the day of Dose 1 administration (Visit 1 of study)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 53
Percentage of participants
  Fever: >=38.0 deg C | 7.7 [2.1 to 18.5] | 18.9 [9.4 to 32.0]
  Fever: >=38.0 deg C to 38.4 deg C | 3.8 [0.5 to 13.2] | 9.4 [3.1 to 20.7]
  Fever: >38.4 deg C to 38.9 deg C | 1.9 [0.0 to 10.3] | 7.5 [2.1 to 18.2]
  Fever: >38.9 deg C to 40.0 deg C | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.1]
  Fever: >40.0 deg C | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Decreased appetite: Any | 40.4 [27.0 to 54.9] | 34.0 [21.5 to 48.3]
  Decreased appetite: Mild | 17.3 [8.2 to 30.3] | 15.1 [6.7 to 27.6]
  Decreased appetite: Moderate | 21.2 [11.1 to 34.7] | 18.9 [9.4 to 32.0]
  Decreased appetite: Severe | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.7]
  Decreased appetite: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Drowsiness: Any | 53.8 [39.5 to 67.8] | 50.9 [36.8 to 64.9]
  Drowsiness: Mild | 42.3 [28.7 to 56.8] | 32.1 [19.9 to 46.3]
  Drowsiness: Moderate | 9.6 [3.2 to 21.0] | 17.0 [8.1 to 29.8]
  Drowsiness: Severe | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.1]
  Drowsiness: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]
  Irritability: Any | 73.1 [59.0 to 84.4] | 67.9 [53.7 to 80.1]
  Irritability: Mild | 23.1 [12.5 to 36.8] | 26.4 [15.3 to 40.3]
  Irritability: Moderate | 42.3 [28.7 to 56.8] | 37.7 [24.8 to 52.1]
  Irritability: Severe | 7.7 [2.1 to 18.5] | 3.8 [0.5 to 13.0]
  Irritability: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.7]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Fever (oral temperature >= 38 degC) was categorized as >=38.0-38.4 degC, >38.4-38.9 degC, >38.9-40.0 degC and >40.0 degC. Decreased appetite was graded as mild: decreased interest in eating, moderate: decreased oral intake, severe: refusal to feed. Drowsiness was graded as mild: increased/prolonged sleeping bouts, moderate: slightly subdued, interfered daily activity, severe: disabled, not interested in daily activity. Irritability was graded as mild: easily consolable, moderate: required increased attention, severe: inconsolable, crying couldn't be comforted. Grade 4 decreased appetite, drowsiness and irritability events led to emergency room visit or hospitalization and were classified by investigator/medically qualified person. Any systemic event: any fever, decreased appetite, drowsiness, irritability.
Time Frame: Day 1 through Day 7, where Day 1 is the day of Dose 2 administration (Visit 3 of study)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 51
Percentage of participants
  Fever: >=38.0 deg C | 13.5 [5.6 to 25.8] | 15.7 [7.0 to 28.6]
  Fever: >=38.0 deg C to 38.4 deg C | 9.6 [3.2 to 21.0] | 7.8 [2.2 to 18.9]
  Fever: >38.4 deg C to 38.9 deg C | 1.9 [0.0 to 10.3] | 2.0 [0.0 to 10.4]
  Fever: >38.9 deg C to 40.0 deg C | 1.9 [0.0 to 10.3] | 5.9 [1.2 to 16.2]
  Fever: >40.0 deg C | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Decreased appetite: Any | 23.1 [12.5 to 36.8] | 31.4 [19.1 to 45.9]
  Decreased appetite: Mild | 7.7 [2.1 to 18.5] | 7.8 [2.2 to 18.9]
  Decreased appetite: Moderate | 15.4 [6.9 to 28.1] | 23.5 [12.8 to 37.5]
  Decreased appetite: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Decreased appetite: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Drowsiness: Any | 30.8 [18.7 to 45.1] | 31.4 [19.1 to 45.9]
  Drowsiness: Mild | 17.3 [8.2 to 30.3] | 25.5 [14.3 to 39.6]
  Drowsiness: Moderate | 11.5 [4.4 to 23.4] | 5.9 [1.2 to 16.2]
  Drowsiness: Severe | 1.9 [0.0 to 10.3] | 0 [0.0 to 7.0]
  Drowsiness: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]
  Irritability: Any | 53.8 [39.5 to 67.8] | 49.0 [34.8 to 63.4]
  Irritability: Mild | 21.2 [11.1 to 34.7] | 19.6 [9.8 to 33.1]
  Irritability: Moderate | 30.8 [18.7 to 45.1] | 29.4 [17.5 to 43.8]
  Irritability: Severe | 1.9 [0.0 to 10.3] | 0 [0.0 to 7.0]
  Irritability: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 7.0]

5. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 Through 1 Month After Dose 2
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Results excluded local reactions and systemic events data.
Time Frame: From Dose 1 through 1 month after Dose 2 [up to approximately 3.7 months]
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 53
Percentage of participants | 84.6 [71.9 to 93.1] | 75.5 [61.7 to 86.2]

6. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 Through 1 Month After Dose 2
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic; other situations as judged by investigator.
Time Frame: From Dose 1 through 1 month after Dose 2 [up to approximately 3.7 months]
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 52 | 53
Percentage of participants | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.1]

7. Secondary Outcome: Geometric Mean Concentration (GMCs) of Pneumococcal Immunoglobulin G (IgG) at 1 Month After Dose 1
Description: GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the student t distribution).
Time Frame: 1 month after Dose 1
Population: Dose 1 evaluable immunogenicity population included all participants who were eligible and randomized, received the study intervention to which they were randomized, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 1, and had no other major protocol deviations as determined by the clinician up to the 1-month post-Dose 1 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram/milliliter (mcg/mL)
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 50 | 49
Microgram/milliliter (mcg/mL) | 7.53 [5.68 to 9.99] | 5.73 [4.51 to 7.29]

8. Secondary Outcome: GMCs of Pneumococcal IgG at 1 Month After Dose 2
Description: as for outcome 7
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population included all participants who were eligible and randomized, received both doses of study intervention to which they were randomly assigned, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 2, and had no other major protocol deviations as determined by the clinician up to the 1-month post-Dose 2 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram/milliliter (mcg/mL)
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 50 | 48
Microgram/milliliter (mcg/mL) | 17.41 [13.90 to 21.79] | 8.08 [6.42 to 10.16]

9. Secondary Outcome: Percentage of Participants With Predefined IgG Concentrations at 1 Month After Dose 1
Description: Predefined IgG concentrations was >= 0.35 micrograms per milliliter (mcg/mL).
Time Frame: 1 month after Dose 1
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 50 | 49
Percentage of participants | 98.0 [89.4 to 99.9] | 100.0 [92.7 to 100.0]

10. Secondary Outcome: Percentage of Participants With Predefined IgG Concentrations at 1 Month After Dose 2
Description: Predefined level of IgG concentrations was >= 0.35 mcg/mL.
Time Frame: 1 month after Dose 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 50 | 48
Percentage of participants | 100.0 [92.9 to 100.0] | 100.0 [92.6 to 100.0]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFRs) of Pneumococcal IgG From Before Dose 1 to 1 Month After Dose 1
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student-t distribution).
Time Frame: From before Dose 1 to 1 month after Dose 1
Population: Dose 1 evaluable immunogenicity population included all participants who were eligible and randomized, received study intervention to which they were randomized, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 1, and had no other major protocol deviations as determined by clinician up to 1-month post-Dose 1 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 1 evaluable participants with valid result at both timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 46 | 46
Fold rise | 496.7 [316.2 to 780.3] | 306.3 [196.7 to 476.9]

12. Secondary Outcome: GMFRs of Pneumococcal IgG From 1 Month After Dose 1 to 1 Month After Dose 2
Description: as for outcome 11
Time Frame: From 1 month after Dose 1 to 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population included all participants who were eligible, randomized, received both doses of study intervention to which they were randomly assigned, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 2, had no major protocol deviations as determined by clinician up to 1-month post-Dose 2 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 2 evaluable participants with valid result at both timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 48 | 45
Fold rise | 2.4 [1.9 to 2.9] | 1.5 [1.3 to 1.7]

13. Secondary Outcome: Geometric Mean Titer (GMTs) of Pneumococcal Opsonophagocytic Activity (OPA) at 1 Month After Dose 1
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution).
Time Frame: 1 month after Dose 1
Population: Dose 1 evaluable immunogenicity population included all participants who were eligible and randomized, received study intervention to which they were randomized, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 1, and had no other major protocol deviations as determined by clinician up to 1-month post-Dose 1 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 1 evaluable participants with valid OPA titers.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 49 | 48
Titer | 425 [346 to 522] | 447 [363 to 550]

14. Secondary Outcome: GMTs of Pneumococcal OPA at 1 Month After Dose 2
Description: as for outcome 13
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population included all participants who were eligible, randomized, received both doses of study intervention to which they were randomly assigned, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 2, had no major protocol deviations as determined by clinician up to 1-month post-Dose 2 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 2 evaluable participants with valid OPA titers.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 50 | 47
Titer | 645 [538 to 773] | 544 [455 to 650]

15. Secondary Outcome: GMFRs of Pneumococcal OPA From Before Dose 1 to 1 Month After Dose 1
Description: as for outcome 11
Time Frame: From before Dose 1 to 1 month after Dose 1
Population: Dose 1 evaluable immunogenicity population included all participants who were eligible and randomized, received study intervention to which they were randomized, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 1, and had no other major protocol deviations as determined by clinician up to 1-month post-Dose 1 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 1 evaluable participants with valid OPA result at both timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 44 | 45
Fold rise | 40.7 [30.4 to 54.6] | 42.6 [30.3 to 59.9]

16. Secondary Outcome: GMFRs of Pneumococcal OPA From 1 Month After Dose 1 to 1 Month After Dose 2
Description: as for outcome 11
Time Frame: From 1 month after Dose 1 to 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population included all participants who were eligible, randomized, received both doses of study intervention to which they were randomly assigned, had at least 1 valid immunogenicity result within 27 to 56 days, inclusive, after Dose 2, had no major protocol deviations as determined by clinician up to 1-month post-Dose 2 visit. Here, ''Overall Number of Participants Analyzed'' signifies Dose 2 evaluable participants with valid OPA result at both timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | mPnC Candidate | mPnC Control
Number analyzed (Participants) | 47 | 43
Fold rise | 1.5 [1.2 to 1.9] | 1.3 [1.1 to 1.5]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic collection): Within 7 days after Dose 1 and Dose 2; AEs, SAEs and all-cause mortality (non-systematic collection): From Dose 1 through 1 month after Dose 2 [up to approximately 3.7 months]
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | mPnC Candidate | mPnC Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/53
Other Adverse Events (participants affected / at risk) | 51/52 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mPnC Candidate (N=52) | mPnC Control (N=53)
Bronchitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mPnC Candidate (N=52) | mPnC Control (N=53)
Pyrexia (General disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Gastroenteritis (Infections and infestations) | 14 | 12
Nasopharyngitis (Infections and infestations) | 8 | 5
Otitis media (Infections and infestations) | 5 | 4
Rhinitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 24 | 22
Injection site erythema (REDNESS) (General disorders) | 13 | 15
Injection site pain (PAIN) (General disorders) | 16 | 19
Injection site swelling (SWELLING) (General disorders) | 8 | 6
Pyrexia (FEVER) (General disorders) | 8 | 15
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 26 | 25
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 31 | 33
Irritability (IRRITABILITY) (Psychiatric disorders) | 42 | 43
Vomiting (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT06116591/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT06116591/SAP_001.pdf